CLINICAL TRIAL: NCT06751498
Title: The Value of a Renal Artery Perfusion Model Based on Convolutional Neural Network in Predicting Renal Function After Partial Nephrectomy: A Prospective, Single-Center Study
Brief Title: The Value of a Convolutional Neural Network-Based Renal Artery Perfusion Model in Predicting Renal Function After Partial Nephrectomy: A Prospective Study
Status: Recruiting | Type: Observational
Sponsor: Shao Pengfei (Other)
Responsible Party: Sponsor-Investigator, Shao Pengfei, chief physician, The First Affiliated Hospital with Nanjing Medical University
Organization: The First Affiliated Hospital with Nanjing Medical University (Other)
Other Study IDs: 2024-SR-710
Record Dates: First submitted 2024-12-25; First posted 2024-12-30 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Renal Cell Cancer
Keywords: Articicial Intelligence; convolutional neural network; renal arterial perfusion model; partial nephrectomy; fractional renal function
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to develop a CNN-based machine module to predict postoperative fractional renal function in people who are proposed to undergo partial nephrectomy. The main question it aims to answer is:

• Does this machine learning model accurately predict renal function after partial nephrectomy?

DETAILED DESCRIPTION:
This prospective study is conducted to predict postoperative fractional renal function using the perfusion deficit method from a preoperatively established renal arterial perfusion model for people who are proposed to undergo partial nephrectomy. In this study, this prediction method will be compared with the true missing values of renal units on nuclear renal function, eGFR, and CTA. This study aims to evaluate the feasibility of applying the CNN-based model in predicting postoperative renal function after partial nephrectomy and provide high-level clinical evidence for the preoperative integrated diagnostic and treatment process of renal tumors, especially in terms of the functional evaluation.

ELIGIBILITY:
Inclusion Criteria:

* people with stage cT1 renal tumors confirmed by preoperative CT or MR
* people who are proposed to undergoing partial nephrectomy
* localized renal tumors without lymph node and distant metastases as defined by NCCN guidelines
* ECOG score of 0 or 1
* Life expectancy greater than 10 years

Exclusion Criteria:

* people with surgically unresectable lesions
* people with Abnormal preoperative renal function, eGFR(estimated by CKD-EPI)<90ml/min/1.73m2
* people who receive preoperative molecular targeted therapy, immunotherapy, chemotherapy
* people with any contraindications to surgery
* people who convert to radical nephrectomy during surgery
* people who receive molecular targeted therapy, immunotherapy or chemotherapy during the postoperative follow-up period
* people with serious systemic disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: people with localized renal tumors scheduled for partial nephrectomy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
GFR of ipsilateral and contralateral kidneys | 3 months after surgery
volume of ipsilateral kidney | 3 months after surgery

SECONDARY OUTCOMES:
Postoperative total renal function(eGFR) | 24 hours, 1 month, 3 months, 6 months, 1 year after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University (Jiangsu Provincial People's Hospital), Nanjing, Jiangsu, China